CLINICAL TRIAL: NCT00679640
Title: Observational Usage and Efficacy Study of Candesartan in Heart Failure Treatment in France
Acronym: SISTOLA
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Deborah Watts, Astrazeneca
Other Study IDs: NIS-CFR-ATA-2007/1
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-07

CONDITIONS: Heart Failure; Cohort Study
Keywords: candesartan; heart failure; cohort study; France
MeSH Terms: conditions — Heart Failure | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Outpatients to whom candesartan has been initiated for less than 30 days or during the consultation to treat heart failure
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Candesartan — Oral tablets
  Other Names: Atacand

SUMMARY:
The purpose of this study is to describe the way candesartan is used in heart failure treatment in France (treatment initiation and monitoring), treatment stops occurrence and reasons for and patients clinical evolution

ELIGIBILITY:
Inclusion Criteria:

* outpatients to whom candesartan has been initiated for less than 30 days or during the consultation to treat heart failure

Exclusion Criteria:

* patients included in a clinical trial the last 30 days before consultation
* patients unable to answer the questions for linguistic or cognitive reasons
* patients who will be difficult to follow during the one year study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen in outpatient care (private consultation or outpatient hospital consultation) at the baseline visit
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Profile of patients treated with candesartan for heart failure | At inclusion

SECONDARY OUTCOMES:
Percentage of patients taking correctly its treatment : indication, contraindication, drug titration, treatment monitoring | 6 and 12 months after
Percentage of patients stopping its treatment and reasons why | 12 months after
Percentage of hospitalisations due to heart failure and cardiovascular deaths | 12 months after

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Bouee, MD, MSc, Principal Investigator — CEMKA EVAL - Bourg La Reine - France; Luc Hittinger, MD, Prof, Study Chair — Hôpital Henri Mondor - Service de cardiologie - Créteil - France
Locations (103):
- France (103):
  - Research Site, Mulhouse, Alsace
  - Research Site, Bordeaux, Aquitaine Nord
  - Research Site, Dax, Aquitaine Sud
  - Research Site, Saint-Jean-de-Luz, Aquitaine Sud
  - Research Site, Tarbes, Aquitaine Sud
  - Research Site, Arras, Artois
  - Research Site, Béthune, Artois
  - Research Site, Besançon, Aube Franche Comte
  - Research Site, Langres, Aube Franche Comte
  - Research Site, Vesoul, Aube Franche Comte
  - Research Site, Clermont-Ferrand, Auvergne Stephanois
  - Research Site, Saint-Chamond, Auvergne Stephanois
  - Research Site, Saint-Etienne, Auvergne Stephanois
  - Research Site, Caen, Basse Normandie
  - Research Site, Granville, Basse Normandie
  - Research Site, Mayenne, Basse Normandie
  - Research Site, Saint-Martin-d'Aubigny, Basse Normandie
  - Research Site, Valognes, Basse Normandie
  - Research Site, Dijon, Bourgogne-Franche-Comté
  - Research Site, Dole, Bourgogne-Franche-Comté
  - Research Site, Paray-le-Monial, Bourgogne-Franche-Comté
  - Research Site, Semur-en-Auxois, Bourgogne-Franche-Comté
  - Research Site, Lannion, Bretagne Nord
  - Research Site, Rennes, Bretagne Nord
  - Research Site, Morlaix, Bretagne Sud
  - Research Site, Bry-sur-Marne, Brie
  - Research Site, Meaux, Brie
  - Research Site, Savigny-sur-Orge, Brie
  - Research Site, Béziers, Catalogne
  - Research Site, Perpignan, Catalogne
  - Research Site, Sète, Catalogne
  - Research Site, Épernay, Champagne Ardennes
  - Research Site, Château-d'Olonne, Charente
  - Research Site, Niort, Charente
  - Research Site, Poitiers, Charente
  - Research Site, Royan, Charente
  - Research Site, Annecy-le-Vieux, Dauphine
  - Research Site, Annemasse, Dauphine
  - Research Site, Sallanches, Dauphine
  - Research Site, Nice, Esterel
  - Research Site, Saint-Raphaël, Esterel
  - Research Site, Hazebrouck, Flandres
  - Research Site, Lille, Flandres
  - Research Site, Wattrelos, Flandres
  - Research Site, Castelsarrasin, Gascogne
  - Research Site, Montauban, Gascogne
  - Research Site, Périgueux, Gascogne
  - Research Site, Rouen, Haute Normandie
  - Research Site, Boulogne-Billancourt, Hauts de Seine
  - Research Site, Arles, Languedoc
  - Research Site, Montpellier, Languedoc
  - Research Site, Nîmes, Languedoc
  - Research Site, Rodez, Languedoc
  - Research Site, Villefranche-de-Rouergue, Languedoc
  - Research Site, Limoges, Limousin
  - Research Site, Saint-Amand-Montrond, Limousin
  - Research Site, Saint-Yrieix-la-Perche, Limousin
  - Research Site, Nancy, Lorraine
  - Research Site, Saint-Avold, Lorraine
  - Research Site, Bourgoin, Lyonnais
  - Research Site, Bron, Lyonnais
  - Research Site, Gleizé, Lyonnais
  - Research Site, Lyon, Lyonnais
  - Research Site, Rillieux-la-Pape, Lyonnais
  - Research Site, Cogolin, Maures Corse
  - Research Site, Hyères, Maures Corse
  - Research Site, Toulon, Maures Corse
  - Research Site, Castanet-Tolosan, Midi Pyrenees
  - Research Site, Muret, Midi Pyrenees
  - Research Site, Paris, Paris Centre
  - Research Site, Aulnay-sous-Bois, Paris Nord Est
  - Research Site, Montfermeil, Paris Nord Est
  - Research Site, Montreuil, Paris Nord Est
  - Research Site, Châteaubriant, Pays de Loire
  - Research Site, Nantes, Pays de Loire
  - Research Site, Amiens, Picardie
  - Research Site, Condé-sur-l'Escaut, Picardie
  - Research Site, Valenciennes, Picardie
  - Research Site, Allauch, Provence-Alpes-Côte d'Azur Region
  - Research Site, Marseille, Provence-Alpes-Côte d'Azur Region
  - Research Site, Rognac, Provence-Alpes-Côte d'Azur Region
  - Research Site, Salon-de-Provence, Provence-Alpes-Côte d'Azur Region
  - Research Site, La Source, Sologne
  - Research Site, Montargis, Sologne
  - Research Site, Orléans, Sologne
  - Research Site, Tonnerre, Sologne
  - Research Site, Arpajon, Touraine
  - Research Site, Chambray-lès-Tours, Touraine
  - Research Site, Tours, Touraine
  - Research Site, Villiers-sur-Orge, Touraine
  - Research Site, Apt, Vallee Du Rhone
  - Research Site, Châteaurenard, Vallee Du Rhone
  - Research Site, Gap, Vallee Du Rhone
  - Research Site, Beauchamp, Vexin
  - Research Site, Beauvais, Vexin
  - Research Site, Cergy, Vexin
  - Research Site, Chelles, Vexin
  - Research Site, Creil, Vexin
  - Research Site, Pontoise, Vexin
  - Research Site, Sarcelles, Vexin
  - Research Site, Évecquemont, Yvelines
  - Research Site, Gennevilliers, Yvelines
  - Research Site, Maisons-Laffitte, Yvelines